CLINICAL TRIAL: NCT05148845
Title: Open-label, Single-arm Phase 3B Implementation Study to Evaluate the Effectiveness of the Homologous Boostof Ad26.COV2.S COVID-19 Vaccine Following the Prime Dose Among Sisonke Participants in South Africa(VAC31518COV30XX)
Brief Title: Sisonke 2 - A COVID-19 Vaccine Boost Open Label Study.
Acronym: Sisonke Boost
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: National Department of Health of South Africa (Unknown); National Institute of Communicable Diseases - NICD (Unknown); KwaZulu-Natal Research Innovation and Sequencing Platform - KRISP (Unknown); Fred Hutchinson Cancer Center (Other); Hutchinson Center Research Institute of South Africa (HCRISA) (Unknown); Janssen Vaccines & Prevention B.V. (Industry); Bio Analytical Research Corporation (Industry); Dis-Chem Pharmacy (Unknown); BioVac (Unknown); Biocair (Unknown); Right to Care (Other); Clinical Laboratory Services (Other); Institute of Infectious Disease and Molecular Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Sisonke Boost Open Label Study
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2021-12

CONDITIONS: SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm phase 3B vaccine implementation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Booster vaccine — To evaluate the effectiveness and safety of the single dose Ad26.COV2.S (Jansen) COVID-19 vaccine plus a homologous boost with Ad26.COV2.S (Janssen) COVID-19 vaccine among Sisonke participants as compared to unboosted Sisonke participants
  In addition we will continue to evaluate VE of the Sisonke Boost compared to:
  i) Vaccinated populations pre boosts ii) Unvaccinated populations in South Africa.

SUMMARY:
To evaluate the effectiveness of the single dose Ad26.COV2.S COVID-19 vaccine plus a homologous boostwith Ad26.COV2.S COVID-19 vaccine among Sisonke participants as compared to unboosted Sisonkeparticipants; vaccinated; and unvaccinated populations in South Africa

DETAILED DESCRIPTION:
Purpose To evaluate the effectiveness and safety of the single dose Ad26.COV2.S (Jansen) COVID-19 vaccine plus a homologous boost with Ad26.COV2.S (Janssen) COVID-19 vaccine among Sisonke participants as compared to unboosted Sisonke participants

In addition the investigators will continue to evaluate VE of the Sisonke Boost compared to:

i) Vaccinated populations pre boosts ii) Unvaccinated populations in South Africa.

Study design Open-label, single-arm phase 3B vaccine implementation study

Rationale South Africa is severely affected by the global COVID-19 epidemic, and following the initial prime vaccination among HCWs in the first 4 months of 2021. New data has demonstrated the safety and effectiveness of a booster dose given two months or more after the initial Ad26.COV2.S. This provides the rationale and feasibility for the evaluation of a homologous booster vaccine dose to the cohort of vaccinated Sisonke participants to inform the larger vaccine rollout.

Study participants Sisonke participants age 18 and over working in the South African public and private health care sector (approx N=500 000) who were enrolled in Sisonke and have not subsequently had a further booster vaccine dose.

Study sites Department of Health Vaccine Administration Sites across South Africa supported by the Sisonke (Together) (VAC31518COV3012) Trial Research Site Investigators and Study Staff

Study duration Participants will receive a homologous Ad26.COV2.S (Janssen) booster dose of vaccine at least 6 months post the prime vaccination. The investigators will monitor outcomes utilising the DATCOV surveillance system and NHLS/NICD SARS COV-2 testing databases for up to 2 years post initial vaccination.

Study products Ad26.COV2.S by Janssen administered as a single dose followed by a single booster injection.

Primary objectives • To assess the effectiveness of Ad26.COV2.S vaccine as a homologous boost on severe COVID, hospitalizations and deaths in Sisonke participants as compared with the unboosted Sisonke populations.

Secondary objectives To assess the effectiveness of Ad26.COV2.S vaccine as a homologous boost on severe COVID, hospitalizations and deaths in Sisonke participants as compared vaccinated and unvaccinated populations of essential workers in South Africa.

* To estimate the incidence of symptomatic SARS CoV-2 infections in Sisonke participants following a boost compared with the unboosted Sisonke populations and general vaccinated and unvaccinated population in South Africa
* To estimate booster dose uptake among Sisonke participants in South Africa
* To monitor the genetic diversity of breakthrough SARS CoV-2 infections.
* To monitor safety in the case of homologous boosts in Sisonke participants.

ELIGIBILITY:
Inclusion Criteria

* Age 18 and older
* All Sisonke participants
* Received a priming Ad26.SARS.COV.2.S vaccination as part of the Sisonke study at least 6 months prior
* Participants who are pregnant or report breastfeeding at the time of enrolment may be included.
* Willingness and ability to comply with vaccination plan and other study procedures.
* Capable of giving electronic or personal signed informed consent as described in Appendix 5, which includes compliance with the requirements in this protocol.

Exclusion Criteria:

* Participants who have received boosting vaccination through other means.
* Any significant acute or chronic medical condition, situation or circumstance that in the opinion of the PI/designee makes the participant unsuitable for participation in the study, or jeopardises the safety or rights of the participant
* Current participation in any other research studies that would interfere with the objectives of this study. The determination of whether participation in another study would be exclusionary for a given participant will be made by the PI/designee.
* Participants with a history of heparin-induced thrombocytopenia or TTS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500000 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of Ad26.COV2.S (Janssen) boost vaccine on severe COVID, hospitalizations and deaths in Sisonke participants as compared to unboosted Sisonke participants (single Ad26 vaccine only) | 24 Months
  Rates of hospitalizations and deaths among boosted Sisonke participants versus unboosted Sisonke participants and unvaccinated populations in South Africa

SECONDARY OUTCOMES:
To assess the effectiveness of Ad26.COV2.S (Janssen) boost vaccine on severe COVID, hospitalizations and deaths in Sisonke participants as compared to the vaccinated and unvaccinated populations (no vaccination) in South Africa. | 24 Months
  Rates of hospitalizations and deaths among boosted Sisonke participants versus unboosted vaccinated and unvaccinated populations in South Africa
To estimate the incidence of symptomatic SARS CoV-2 infections among boosted Sisonke ppts. | 24 months
  Incidence rate of SARS CoV-2 infection as indicated by self-report and validation in national laboratory records.
  Rates of severe disease in Sisonke participants who are found to be RT-PCR positive at any time up to 2 years post prime vaccination
To monitor the genetic diversity of breakthrough SARS CoV-2 infections | 24 Months
  Genetic diversity of breakthrough infection virus as determined by whole genome sequencing. This will be recovered from national laboratories.
To estimate booster vaccine uptake among Sisonke participants in South Africa | 24 Months
  Proportion of Sisonke participants approached for study participation taking part in the boost study and receiving the booster vaccine
To monitor safety in homologous boosts | 24 Months
  All SAEs and events of special interest will be collected and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, MBChB, Principal Investigator — Non-Executive Director
Locations (31):
- South Africa (31):
  - Nelson Mandela Academic Clinical Research Unit (NeMACRU), Mthatha, Eastern Cape
  - PHOENIX Pharma Pty Ltd, Port Elizabeth, Eastern Cape
  - Josha Research, Bloemfontein, Free State
  - Perinatal HIV Research Unit (PHRU), SOWETO, Johannesburg, Gauteng
  - Clinical HIV Research Unit (CHRU),, Johannesburg, Gauteng
  - MeCRU Clinical Research Unit, Pretoria, Gauteng
  - Setshaba Research Centre,, Pretoria, Gauteng
  - The Aurum Institute Clinical Research Centre, Pretoria, Pretoria, Gauteng
  - Ndlovu Research Centre, Pretoria, Gauteng
  - The Aurum Institute: Tembisa Clinical Research Centre, Johannesburg, Gauteng - South
  - Perinatal HIV Research Unit Kliptown, Johannesburg, Gauteng - South
  - Botha's Hill Clinical Research Site, Bothas Hill, KwaZulu-Natal
  - CAPRISA eThekwini Clinical Research Site, Dr, Durban, KwaZulu-Natal
  - Chatsworth Clinical Research Site, Durban, KwaZulu-Natal
  - CAPRISA Vulindlela Clinical Research Site, Dr Disebo Makhaza, Durban, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic, Ladysmith, KwaZulu-Natal
  - Tongaat Clinical Research Site, Dr, Tongaat, KwaZulu-Natal
  - Mzansi Ethical Research Centre, Middleburg, Mpumalanga
  - The Aurum Institute Klerksdorp Clinical Research Centre, Klerksdorp, North West
  - TASK Applied Science, Delft Day Hospital Premises, Cape Town, Western Cape
  - TASK Applied Science, Dr Ivans Toms Clinic Premises, Cape Town, Western Cape
  - FAMCRU (Family Clinical Research Unit),, Cape Town, Western Cape
  - TASK Applied Science, Brooklyn Chest Hospital Premises, Cape Town, Western Cape
  - TASK Central, Cape Town, Western Cape
  - TASK Clinical Research Centre, Cape Town, Western Cape
  - Emavundleni Research Centre, Cape Town, Western Cape
  - Desmond Tutu Health Foundation CTU J52 Old Main Building Groote SchuurHospital, Cape Town, Western Cape
  - TASK Eden, George, Western Cape
  - South African Vaccine Initiative (SATVI), Worcester, Western Cape
  - Desmond Tutu Health Foundation - Masiphumelele Research Office, Cape Town
  - The Aurum Institute: Rustenburg Clinical Research Centre, Dr Lawrence, Rustenburg

IPD SHARING:
Plan to Share IPD: Yes
All study team scientists will disseminate the trial results as broadly as possible. Data will be shared with JNJ prior to release to the public. The study data will be published consistent with normal scientific practices.
  The results from this research may also be disseminated through presentations at scientific institutions/ meetings, and/or publication in scientific journals. All publications will be uploaded to a publication repository. After sharing the results with study participants, they will be presented to communities from which participants are recruited, following Good Participatory Practice guidelines. The results will also be shared with global and local policy makers. Summary results of the trial will be made publicly available through the clinical trial registry. Any datasets used for analysis in publications can be requested by investigators via an online request to the organisation. Measures will be taken to protect identifiable information in the datasets
Supporting Information: CSR
Time Frame: Within 12 months of completion of study
Access Criteria: on request
URL: https://www.samrc.ac.za

REFERENCES:
- [Derived] Takalani A, Robinson M, Jonas P, Bodenstein A, Sambo V, Jacobson B, Louw V, Opie J, Peter J, Rowji P, Seocharan I, Reddy T, Yende-Zuma N, Khutho K, Sanne I, Bekker LG, Gray G, Garrett N, Goga A; Sisonke Study Team. Safety of a second homologous Ad26.COV2.S vaccine among healthcare workers in the phase 3b implementation Sisonke study in South Africa. Vaccine. 2024 Feb 27;42(6):1195-1199. doi: 10.1016/j.vaccine.2024.01.066. Epub 2024 Jan 25. PMID 38278629